CLINICAL TRIAL: NCT03655925
Title: Plasma Levels of Human Leucocyte Antigen G in Patients With Chronic Heart Failure
Brief Title: Human Leucocyte Antigen G and Chronic Heart Failure
Status: Completed | Type: Observational
Sponsor: Piera Boschetto (Other)
Responsible Party: Sponsor-Investigator, Piera Boschetto, Professor, University Hospital of Ferrara
Organization: University Hospital of Ferrara (Other)
Other Study IDs: 170687
Record Dates: First submitted 2018-07-25; First posted 2018-08-31 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Chronic Heart Failure (CHF): Entire cohort/ Patients with recent diagnosis of chronic heart failure as defined by the guidelines of the European Society of Cardiology (ESC) and with cardiac ejection fraction <40
  Interventions: Diagnostic Test: plasmatic HLA-G

INTERVENTIONS:
Diagnostic Test: plasmatic HLA-G — plasmatic HLA-G by blood sample

SUMMARY:
The Human leukocyte antigen G (HLA-G) is a non-classical, major histocompatibility complex class I (MHC-I) protein that modulates the immune response, inhibiting it in most cases. Physiologically expressed in the cells of some tissues, it increases in inflammatory reactions. Inflammation appears to play an important role in the development of chronic heart failure. This study aims to evaluate the levels of soluble HLA-G in patients with heart failure and to investigate the relationships between HLA-G and other clinical-functional parameters of the disease. Investigators hypothesize that the plasma levels of HLA-G could correlate with the clinical status of heart failure and could provide indications on patient's prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recent diagnosis of chronic heart failure as defined by the guidelines of the European Society of Cardiology (ESC) and with cardiac ejection fraction <40.
* Clinical stability in the previous month prior to recruitment.
* Absence of coexisting autoimmune diseases.

Exclusion Criteria:

* Subjects with over one year chronic heart failure diagnosis and in clinical stability for less than 1 month.
* Presence of autoimmune diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 40 subjects with chronic stable heart failure with ejection fraction <40, diagnosed according to the European Society of Cardiology Guidelines
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
To measure plasma levels of soluble Human Leucocyte Antigen G (HLA-G) in patients with chronic heart failure (CHF) | Collection of whole blood at baseline, at 6 and 12 months from baseline
  To measure the plasmatic levels of HLA-G in patients with stable chronic heart failure at baseline. To assess possible changes in HLA-G levels, due to CHF exacerbations, at 6 and 12 months from baseline
To measure the polymorphisms of Human Leucocyte Antigen G (HLA-G) gene | Collection of whole blood at baseline
  To analyze the polymorphisms (Insertion/Deletion 14 pb and 3142 C>G) of the HLA-G gene in patients with chronic heart failure (CHF) at baseline

SECONDARY OUTCOMES:
To correlate the plasma levels of HLA-G with clinical-functional parameters of the chronic heart failure (CHF) in patients with CHF | At baseline and after 12 months
  To correlate plasma levels of HLA-G with Brain Natriuretic Peptide (BNP) and left ventricle ejection fraction at baseline and at 12 months from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Sciences/ Medicine of Public Health, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alegre E, Rizzo R, Bortolotti D, Fernandez-Landazuri S, Fainardi E, Gonzalez A. Some basic aspects of HLA-G biology. J Immunol Res. 2014;2014:657625. doi: 10.1155/2014/657625. Epub 2014 Apr 9. PMID 24818168
- [Background] Almasood A, Sheshgiri R, Joseph JM, Rao V, Kamali M, Tumiati L, Ross HJ, Delgado DH. Human leukocyte antigen-G is upregulated in heart failure patients: a potential novel biomarker. Hum Immunol. 2011 Nov;72(11):1064-7. doi: 10.1016/j.humimm.2011.08.016. Epub 2011 Sep 1. PMID 21925559